CLINICAL TRIAL: NCT07371416
Title: Clinical Outcomes of Immature Teeth Treated With Regenerative Endodontic Procedures Using Intracanal Delivery of Omega-3 Fatty Acids
Brief Title: Regenerative Root Canal Treatment of Immature Teeth Using Omega-3 Fatty Acids
Acronym: Regeneration
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MDP.25.04.8
Record Dates: First submitted 2026-01-09; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Immature Permanent Teeth With Open Apex; Pulp Necrosis
Keywords: Regeneration; Immature Permanent Teeth
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — Docosahexaenoic Acids; Calcium Hydroxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 ( Control ) : Traditional induced bleeding technique (Other): A sterile K-file will be inserted 2 mm beyond the canal terminus to induce bleeding and blood clots inside the canal. The canal orifice which is located in the cervical part of the root canal, measuring 2-3 mm, will be sealed using a white mineral trioxide aggregate (MTA) orifice plug. Then, the access cavity will be sealed using bulk-fill flow composite
  Interventions: Drug: Calcium Hydroxide (Ca(OH)2)
- Group 2: Induced bleeding technique with application of Omega-3 Fatty Acids (Other): The procedure will be identical to that of the first group, except that the ω-3 PUFAs (prepared at the Department of Pharmacognosy, Faculty of Pharmacy, Mansoura University) will be delivered into the root canal during the revascularization procedure. The canal orifice will be sealed in the same manner as in the first group.
  Interventions: Drug: Omega -3 fatty acids; Drug: Calcium Hydroxide (Ca(OH)2)

INTERVENTIONS:
Drug: Omega -3 fatty acids — used within the Regenerative procedures
  Other Names: Omega-3 PUFAs
  Arms: Group 2: Induced bleeding technique with application of Omega-3 Fatty Acids
Drug: Calcium Hydroxide (Ca(OH)2) — Used as intracanal medicament
  Other Names: Ca(OH)2

SUMMARY:
This clinical study will be conducted to evaluate the effect of using intracanal Omega-3 Fatty acids during revascularization of necrotic immature teeth compared to the traditional induced bleeding technique.

DETAILED DESCRIPTION:
Immature permanent teeth with pulp necrosis have thin, fragile dentinal walls, making conventional endodontic sealing techniques challenging. Regenerative endodontics (RE) offers a biologically based alternative that enables continued root development, apical closure, and potential restoration of vitality through approaches such as tissue engineering and revascularization. These procedures rely heavily on the survival and differentiation of stem cells from the apical papilla, even in the presence of infection.

Inflammation plays a pivotal role in RE, influencing both healing and regenerative outcomes. Specialized pro-resolving mediators (SPMs), derived from omega-3 and omega-6 fatty acids, actively resolve inflammation and promote tissue regeneration. Among them, Resolvin E1 (RvE1), derived from EPA, has shown potent anti-inflammatory and pro-regenerative effects, including inhibition of leukocyte infiltration and enhancement of dental pulp stem cell recruitment. Experimental studies demonstrated that intracanal RvE1 reduced periapical inflammation and promoted root development more effectively than traditional intracanal medicaments.

Omega-3 polyunsaturated fatty acids (ω-3 PUFAs), particularly EPA and DHA, have been widely studied in dentistry for their anti-inflammatory and regenerative properties. Evidence from animal studies and clinical trials indicates that ω-3 PUFAs reduce inflammatory mediators, suppress bone resorption, enhance new bone formation, and support stem cell proliferation and differentiation, even under inflammatory conditions. Clinically, ω-3 PUFAs have shown benefits in periodontal therapy, oral mucositis, and other inflammatory oral diseases.

Despite these promising findings, clinical evidence supporting the use of ω-3 PUFAs in endodontics remains limited. Further research is needed to evaluate their role in regenerative endodontic procedures, particularly in necrotic immature teeth where mechanical disinfection is restricted and preservation of apical stem cells is critical. The proposed hypothesis is that ω-3 PUFAs may enhance regenerative endodontic outcomes by modulating inflammation and supporting tissue regeneration.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 6 and 28 years.
* Systemically healthy patients with no history of systemic diseases.
* Patients with necrotic immature permanent teeth due to trauma and/or caries.
* Preoperative radiographic evidence of incomplete root formation.
* Wide apical foramen (apical diameter ≥ 1 mm).
* Thin dentinal walls on preoperative radiographs.

Exclusion Criteria:

* Patients with known allergy to any of the drugs used in the study.
* Patients with systemic diseases or medically compromised conditions.
* Grossly decayed or fractured teeth requiring post and core restorations.
* Presence of draining sinus tract.
* Presence of periodontal pockets.
* Radiographic evidence of external or internal root resorption.
* Patients with a history of major surgeries (e.g., cardiac surgery, kidney transplantation).
* Patients undergoing hemodialysis.

Ages: 6 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Increase in Root Length | 12 months
  Radiographic increase in root length (Millimeters (mm))
Increase in Dentinal Wall Thickness | 12 months
  Radiographic increase in dentinal wall thickness measured using digital image analysis ( Millimeters (mm) )
Periapical Bone Formation | 12 months
  Radiographic evidence of periapical bone formation

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt